CLINICAL TRIAL: NCT04624321
Title: Study to Evaluate the Digital Health and Lifestyle Tool Developed at the University of Gothenburg
Brief Title: Assessment of the Health and Lifestyle Tool
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Health1
Record Dates: First submitted 2020-10-30; First posted 2020-11-10 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Health

STUDY DESIGN:
Intervention Model Description: The study has an initial 3-month randomization phase with two parallel arms, one randomized to access the lifestyle tool and one randomized to a wait list on usual care. After that 3-month period, all participants will get access to the tool, independent of previous randomization assignment, and are followed over three years in an open-label observation period where changes to HbA1c and secondary variables are compared against matched controls on usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to tool (Experimental): Access to the digital tool. They use the tool at their own and do the different themes that are available. They are recommended to use it at least every other week.
  Interventions: Behavioral: Health and lifestyle tool
- Usual care (Placebo Comparator): They are followed by their ordinary healthcare provider.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Health and lifestyle tool — Health and lifestyle tool used online
  Arms: Access to tool
Other: Usual care — Usual care at ordinary healthcare provider
  Arms: Usual care

SUMMARY:
The overall aim of the study is to evaluate a digital lifestyle intervention that has been developed in an academic setting at the University of Gothenburg, Sweden. The tool is based on self-affirmation theory and has large emphasis on self-reflection to enable sustainable lifestyle changes. The effects of the tool on HbA1c, reflecting long-term blood glucose, will be evaluated in patients with type 2 diabetes. The study will contain two phases. The study consists of a three-month period in which participants are randomly assigned to usual care or access to the intervention tool, followed by an open-label three-year observation period during which participants have access to the tool in addition to ordinary healthcare and are compared with matched controls on usual care.

DETAILED DESCRIPTION:
Considerable evidence suggest that lifestyle interventions can prevent or delay the onset of type 2 diabetes, and self-care behaviors largely determine HbA1c. Modifiable lifestyle factors have been established as key drivers of disease onset, progression, and prognosis, motivating the use of "lifestyle as medicine". Despite this, a substantial number of patients with type 2 diabetes (T2D) have difficulties attaining adequate glycemic control.

Lifestyle interventions are often complex and difficult to implement on a large scale. Digital health interventions are increasingly incorporated into diabetes care, and have the potential to improve both behavioral and clinical outcomes on a broad basis. However, low levels of uptake, reduced user engagement over time, and low acceptance among patients, raise concerns about their effectiveness. Knowledge on how to design interventions aimed at inducing change by promoting motivation and personal engagement, as well as a better understanding of patient interaction with digital health interventions, could help overcome these challenges and inform the development of a novel and effective health support.

The objective or this study is to evaluate a new web-based tool, developed at the University Gothenburg, Sweden, that aims to support patient autonomy and motivation to make sustainable lifestyle changes.

The investigators will test the hypothesis that users of the tool get improved HbA1c relative to baseline as compared with controls on usual care.

Overall study design The study is an investigator-initiated single-center study conducted at Skåne University Hospital, Sweden, and will follow participants over three years.

Participants with T2D will be recruited by sending letters with study information to patients in the ANDIS (All New Diabetics In Scania) registry in Sweden or by advertisements. If HbA1c is 52 mmol/mol or above participants are included and attend study visits every three months during the first year and every sixth month during the following two years for blood sampling and physical examination.

The study has an initial 3-month randomization period. Thereafter, all participants get access to the tool and used it during an open-label observation period of up to three years.

Study procedures All participants receive an email with a link to their personal account on the tool. This email is sent immediately after the initial visit. Via the link participants set a password, complete an initial questionnaire and are then randomized to immediate access the tool or to be on a three-month wait list (1:1 ratio).

The randomization is performed by a web-based system, using a block size of eight. Randomization is unknown to all participants when completing the initial questionnaire and is also unknown to the study personnel at the initial study visit. Thereafter, randomization is non-blinded, i.e. there is full transparency as to who get access to the tool and not.

Those randomized to the wait list receive usual care, which means that participants are followed by their ordinary healthcare provider. Those participants do not receive any information about the tool or its content during the three-month period. Participants who are randomized to wait receive an invitation to a second study visit after three months. Following the visit, an email is sent with a link to complete the questionnaire after which the tool can be accessed.

Study visits Every physical study visit lasts appr. 20 minutes and includes measurements of length and weight, blood pressure, and estimations of fat and muscle mass by bioimpedance. Fasting blood samples are taken for analysis of HbA1c and other cardiometabolic proteins. Participants will not receive any counselling or lifestyle advice at the study visits. Technical problems are referred to the study coordinator, who may also respond to requests to clarify content in a general manner without providing personal advice. Patients are followed by their ordinary physician throughout the study, i.e. the tool is provided on top of ordinary anti-diabetic treatment and healthcare contacts.

The intervention The tool is web-based and used via a computer or mobile phone. It is used at each individual's preferred pace but participants are recommended to login at least every other week. Every round the participants choose a themes (out of appr. 80 possible covering e.g. food, exercise, stress, self-reflection aspects), which takes appr. 15-30 minutes to complete. Participants then reflect on the content and how it could be implemented in daily life. When returning for next round participants are asked to reflect on any changes done since last time. There is no interaction between individual participants.

Statistics As one primary endpoint an intention-to-treat analysis is used to compare HbA1c between the two randomization groups based on data between first and second visit (DeltaHbA1c). Patients lost to follow-up between first and second visit will not be included in the analysis.

The standard deviation of DeltaHbA1c is 6 mmol/mol over 3 months in ANDIS patients with baseline HbA1c at 52 mmol/mol or above. With 80% power at alpha=0.05, 142 participants are needed to each randomization arm to detect a significant difference between the groups, assuming that the true treatment effect of the intervention is 2 mmol/mol over 3 months.

Enrollment will continue until the required number of participants are reached, accounting for those lost to follow-up during the randomization period.

As another primary endpoint, investigators will during the open-label observation period compare DeltaHbA1c at one year relative to baseline between patients using the tool as recommended and matched controls with usual care(1:2 ratio between exposed and controls).

The standard deviation of DeltaHbA1c is 7 mmol/mol over one year (as observed in patients with baseline HbA1c at 52 mmol/mol or above in the ANDIS cohort). With 80% power at alpha=0.05, 24 participants using the tool as recommended and 48 matched controls are needed to detect a significant difference between the groups, assuming that the true treatment effect of the intervention is 5 mmol/mol.

Subanalysis of MOD patients A data-driven cluster analysis of 9,000 diabetes patients has been performed in the ANDIS registry based on six variables measured at diagnosis: GAD antibodies, age, BMI, HbA1c (reflecting long-term blood glucose), HOMA2-B (reflecting insulin secretion) and HOMA2-IR (reflecting insulin resistance). Four clusters of T2D patients were highlighted, each with different characteristics and risk of complications. One of these cluster, MOD (Mild Obesity-related Diabetes), is characterized by high BMI and insulin resistance but relatively well-preserved insulin secretion. It has been suggested that patients with MOD characteristics would benefit particularly from lifestyle changes. The investigators therefore hypothesize that patients with MOD characteristics would benefit particularly well from the intervention. As a subanalysis the investigators will therefore analyse the interaction between MOD/non-MOD subgroup and exposure to the intervention using a linear model with a term for the cluster variable, a term for the exposure to the intervention and an interaction term.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes at or above 35 years of age
* Diagnosis of diabetes mellitus was based on prior documentation or treatment with anti-hyperglycemic medication or diagnosed according to the WHO criteria (random plasma glucose >11.1 mmol/L or fasting glucose >7.0 mmol/L or HbA1C ≥6.5%).
* written informed consent.

Exclusion Criteria:

* type 1 diabetes, MODY or secondary diabetes
* conditions or treatments that in the judgement of the Investigator could affect the study evaluation
* inability to understand written Swedish
* connection with the study team, funders, authorities, universities or other public or private bodies in such a way that specific interests in the study outcomes could be suspected.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of long-term blood glucose concentration measured as glycated hemoglobin at 3 months | 3 months
  Intraindividual change of long-term blood glucose concentration measured as glycated hemoglobin (HbA1c) at 3 months relative to baseline compared between participants with access to the tool and on usual care.
Change of long-term blood glucose concentration measured as glycated hemoglobin at one year | One year of the open-label observation period
  Intraindividual change of long-term blood glucose concentration measured as glycated hemoglobin (HbA1c) at one year relative to baseline between participants who use the tool as recommended and matched controls on usual care

SECONDARY OUTCOMES:
Change of long-term blood glucose concentration measured as glycated hemoglobin at three years | Three years of the open-label observation period
  Intraindividual change of long-term blood glucose concentration measured as glycated hemoglobin (HbA1c) at three years relative to baseline between participants who use the tool as recommended and matched controls on usual care
Body weight | 3 months, 1 year and 3 years
  Body weight between groups
Insulin resistance | 3 months, 1 year and 3 years
  Insulin resistance measured as HOMA-IR
Fasting blood glucose concentration | 3 months, 1 year and 3 years
  Fasting blood glucose concentration between groups
Physical activity in calories per day | 3 years
  Physical activity in calories per day estimated by International Physical activity questionnaire between users of the tool and controls on usual care. Score measures calorie consumption and ranges from 0 to unlimited
Insulin secretion | 1 year and 3 years
  Insulin secretion estimated by HOMA-B

OTHER OUTCOMES:
Change of long-term blood glucose concentration measured as glycated hemoglobin in participants with and without Mild Obesity-related Diabetes, respectively. | 1 year and 3 years
  As a subanalysis we will analyse the effect of the intervention specifically on patients with Mild Obesity-related Diabetes (MOD). This will be analysed by a formal interaction test between MOD and non-MOD participants exposed or not exposed to the intervention by using a linear model with a term for MOD/non-MOD, a term for the exposure/non-exposure to the intervention and an interaction term.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Rosengren, Principal Investigator — Region Skåne
Locations (1):
- Clinical Research Center, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will be shared after deidentification.
Time Frame: Data will be available after publication.
Access Criteria: To researchers who provide a methodologically sound proposal in order to achieve the aims of that proposal. Proposals should be directed by email to internetverktyg@gu.se

REFERENCES:
- [Derived] Salunkhe VA, Sinha N, Ahlqvist E, Prasad RB, Johansson S, Abrahamsson B, Rosengren AH. Digital lifestyle treatment improves long-term metabolic control in type 2 diabetes with different effects in pathophysiological and genetic subgroups. NPJ Digit Med. 2023 Oct 26;6(1):199. doi: 10.1038/s41746-023-00946-0. PMID 37884680
- [Derived] Dwibedi C, Abrahamsson B, Rosengren AH. Effect of Digital Lifestyle Management on Metabolic Control and Quality of Life in Patients with Well-Controlled Type 2 Diabetes. Diabetes Ther. 2022 Mar;13(3):423-439. doi: 10.1007/s13300-022-01214-2. Epub 2022 Feb 12. PMID 35150403